CLINICAL TRIAL: NCT04974580
Title: Young Adult Vaping Cessation: A Randomized Trial Examining Phone Coaching, Text-based Digital Intervention, and Nicotine Replacement Therapy
Brief Title: Research and Innovation to Stop E-cigarette/Vaping in Young Adults
Acronym: (RISE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other); Optum, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth G Klein, Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: GR120236
Record Dates: First submitted 2021-07-02; First posted 2021-07-23 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Nicotine Dependence; E-Cig Use
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial design will be used where all participants receive quitline-delivered phone counseling, and components to be tested are a digital intervention (with text-based cessation and online cessation support) and nicotine replacement therapy (NRT).
Who Masked: Outcomes Assessor
Masking Description: Evaluators are blinded to the study arm assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CoachingOnlyArm (Experimental): Phone Coaching; no Digital Coaching, no NRT: This arm will receive only the two phone counseling calls which all other arms will receive.
  Interventions: Behavioral: Phone Counseling
- DigitalArm (Experimental): Phone Coaching + Digital Coaching; no NRT: This arm will receive digital content (text messages with links to online materials) in addition to to the two phone counseling calls which all arms will receive.
  Interventions: Behavioral: Phone Counseling; Behavioral: Digital Coaching
- CoachingNRTArm (Experimental): Phone Coaching + NRT; no Digital Coaching: This arm will receive Nicotine Replacement Therapy (NRT) in addition to the two phone counseling calls which all arms will receive.
  Interventions: Drug: Nicotine patch; Behavioral: Phone Counseling
- DigitalNRTArm (Experimental): This arm will receive digital content (text messages with links to online materials) AND Nicotine Replacement Therapy (NRT) in addition to the two phone counseling calls which all arms will receive.
  Interventions: Drug: Nicotine patch; Behavioral: Phone Counseling; Behavioral: Digital Coaching

INTERVENTIONS:
Drug: Nicotine patch — NRT will be discussed and dosed by the study quit coach during coaching calls per quitline dosing protocols. NRT treatment will consist of up to an 8 week supply of nicotine patch, gum, and/or lozenge. NRT will be sent in two 4 week shipments. Participants may be dosed for a single form of NRT or combination NRT (patch plus gum or lozenge) based on coach assessment of nicotine use and participant preference.
  Other Names: Nicotine lozenge; Nicotine gum
  Arms: CoachingNRTArm; DigitalNRTArm
Behavioral: Phone Counseling — Participants in all four arms of the study will receive two proactive phone-based behavioral coaching calls for quitting vaping, which will include making a quit plan, learning to cope with urges to vape, and education on strategies for quitting and staying quit. Calls utilize the quitline evidence-based protocol. The first call lasts approximately 20 minutes, the second calls lasts approximately 10 minutes, and participants are encouraged to call in for ad hoc calls if they would like additional support.
Behavioral: Digital Coaching — Intervention descriptionText-based vaping cessation program that utilizes evidence-based content from the quitline tobacco cessation protocol, as well as links directing participants to additional online educational content (brief videos, audio content, quizzes, and educational activities).
  Arms: DigitalArm; DigitalNRTArm

SUMMARY:
The aim of this study is to test intervention components to help young adults quit vaping. A 2x2 factorial design will be used where all participants receive quitline-delivered behavioral phone counseling, and components to be tested are a digital intervention (with text and online cessation support) and nicotine replacement therapy (NRT).

The research questions and hypotheses for this study are:

1. Which components and combinations of intervention yield the greatest success rates for exclusive vaping cessation among young adult exclusive e-cigarette users? H1: The complete condition (NRT + digital) will yield significantly higher rates of cessation compared to the control condition (quitline only).
2. Does 8 weeks of nicotine replacement therapy (NRT) improve initial cessation outcomes relative to no NRT.

   H2: Providing NRT will yield significantly higher quit rates compared to the No NRT condition.
3. Do tailored text-messages and online support during cessation improve initial cessation outcomes relative to no digital content? Are young adult vapers engaged with and satisfied with digital cessation tools? H3: Digital support will yield significantly higher quit rates compared to no digital support.

H4: Higher engagement in digital content will be associated with higher cessation success rates.

DETAILED DESCRIPTION:
The investigators will recruit a national, nonprobability sample of young adults (18-24 year olds) who vape nicotine. All study components will be delivered by phone, mail, online, and mobile device. All participants will receive up to 2 coaching calls and will be randomized to one of four groups: no NRT, no Digital; Digital, no NRT; NRT, no Digital; or NRT and Digital.

Participants (final sample size n = 504) must complete one coaching call to be enrolled in the study. The two coaching calls (approximately 10-20 minutes each) focus on 5 "keys" for quitting: setting a quit date, conquering urges, managing physical withdrawal symptoms (or addressing nicotine replacement needs for the NRT groups), vape-proofing environment, and social supports.

In this real-world trial, coaches will be trained to assess vaping use and dose NRT taking into account use frequency, nicotine level, and participant preference, leveraging quitline standard protocols. Participants may be sent up to 8 weeks (patch, gum, and or lozenge) of product in two shipments. Combination NRT (patch plus gum or lozenge) may be offered.

The digital cessation content includes a text messaging program with links to online education and support materials. The text program will be tailored to a participant's quit stage, and include education, tips, motivational messages, and assessment questions yielding tailored content. The online content (brief videos, audio podcasts, quizzes, etc) can be viewed in small segments via texted links. Participants can also engage with the online content by navigating through lessons or suggested content.

ELIGIBILITY:
Inclusion Criteria:

* Current, regular user of nicotine e-cigarettes (20+ days in the last month)
* Exclusive e-cigarette user (no other tobacco in the last 30 days; or no other tobacco in the last 90 days if smoked 100+ cigarettes or cigarillos in lifetime)
* Interest in quitting in the next 30 days
* Ownership of a smartphone device
* Ability to speak and read English

Exclusion Criteria:

* Pregnant or breastfeeding
* Individuals with schizophrenia or bipolar disorder who do not report that their condition is currently effectively managed
* Individuals who have experienced a heart attack or stroke in the two weeks prior, or who have been diagnosed with rapid/irregular heartbeat or angina in the six months prior to taking the eligibility screener
* Other household members in study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 508 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Klein, PhD, Principal Investigator — Ohio State University College of Public Health
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gentzke AS, Creamer M, Cullen KA, Ambrose BK, Willis G, Jamal A, King BA. Vital Signs: Tobacco Product Use Among Middle and High School Students - United States, 2011-2018. MMWR Morb Mortal Wkly Rep. 2019 Feb 15;68(6):157-164. doi: 10.15585/mmwr.mm6806e1. PMID 30763302
- [Background] Leavens ELS, Stevens EM, Brett EI, Leffingwell TR, Wagener TL. JUUL in school: JUUL electronic cigarette use patterns, reasons for use, and social normative perceptions among college student ever users. Addict Behav. 2019 Dec;99:106047. doi: 10.1016/j.addbeh.2019.106047. Epub 2019 Jul 9. PMID 31442788
- [Background] Graham AL, Jacobs MA, Amato MS. Engagement and 3-Month Outcomes From a Digital E-Cigarette Cessation Program in a Cohort of 27 000 Teens and Young Adults. Nicotine Tob Res. 2020 Apr 21;22(5):859-860. doi: 10.1093/ntr/ntz097. No abstract available. PMID 31197320
- [Background] Brunnemann KD, Hoffmann D. The pH of tobacco smoke. Food Cosmet Toxicol. 1974 Feb;12(1):115-24. doi: 10.1016/0015-6264(74)90327-7. No abstract available. PMID 4459223
- [Background] Buchanan ND, Grimmer JA, Tanwar V, Schwieterman N, Mohler PJ, Wold LE. Cardiovascular risk of electronic cigarettes: a review of preclinical and clinical studies. Cardiovasc Res. 2020 Jan 1;116(1):40-50. doi: 10.1093/cvr/cvz256. PMID 31696222
- [Background] Tanwar V, Adelstein JM, Grimmer JA, Youtz DJ, Katapadi A, Sugar BP, Falvo MJ, Baer LA, Stanford KI, Wold LE. Preconception Exposure to Fine Particulate Matter Leads to Cardiac Dysfunction in Adult Male Offspring. J Am Heart Assoc. 2018 Dec 18;7(24):e010797. doi: 10.1161/JAHA.118.010797. PMID 30561255
- [Background] Tackett AP, Keller-Hamilton B, Smith CE, Hebert ET, Metcalf JP, Queimado L, Stevens EM, Wallace SW, McQuaid EL, Wagener TL. Evaluation of Respiratory Symptoms Among Youth e-Cigarette Users. JAMA Netw Open. 2020 Oct 1;3(10):e2020671. doi: 10.1001/jamanetworkopen.2020.20671. PMID 33048131
- [Background] Rogers JM. Tobacco and pregnancy: overview of exposures and effects. Birth Defects Res C Embryo Today. 2008 Mar;84(1):1-15. doi: 10.1002/bdrc.20119. PMID 18383133
- [Background] Morean ME, Krishnan-Sarin S, S O'Malley S. Assessing nicotine dependence in adolescent E-cigarette users: The 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Nicotine Dependence Item Bank for electronic cigarettes. Drug Alcohol Depend. 2018 Jul 1;188:60-63. doi: 10.1016/j.drugalcdep.2018.03.029. Epub 2018 Apr 26. PMID 29753155
- [Background] Foulds J, Veldheer S, Yingst J, Hrabovsky S, Wilson SJ, Nichols TT, Eissenberg T. Development of a questionnaire for assessing dependence on electronic cigarettes among a large sample of ex-smoking E-cigarette users. Nicotine Tob Res. 2015 Feb;17(2):186-92. doi: 10.1093/ntr/ntu204. Epub 2014 Oct 19. PMID 25332459
- [Derived] Vickerman KA, Carpenter KM, Mullis K, Shoben AB, Nemeth J, Mayers E, Klein EG. Quitline-Based Young Adult Vaping Cessation: A Randomized Clinical Trial Examining NRT and mHealth. Am J Prev Med. 2025 Feb;68(2):366-376. doi: 10.1016/j.amepre.2024.10.019. Epub 2024 Dec 11. PMID 39665734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Started | 134 | 126 | 126 | 122
Completed | 101 | 87 | 96 | 93
Not Completed | 33 | 39 | 30 | 29
Not completed — Lost to Follow-up | 33 | 39 | 30 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm | Total
Number analyzed (Participants) | 134 | 126 | 126 | 122 | 508
Age, Customized [Count of Participants; unit: Participants]
  Age Category: 18-21 years old | 76 | 80 | 71 | 63 | 290
  Age Category: 22-24 years old | 58 | 46 | 55 | 59 | 218
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 97 | 92 | 85 | 88 | 362
  Gender: Male | 34 | 30 | 34 | 28 | 126
  Gender: Transgender female | 0 | 0 | 0 | 1 | 1
  Gender: Transgender male | 2 | 2 | 3 | 3 | 10
  Gender: Other identity | 1 | 2 | 4 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing race/ethnicity data on one participant (due to not answering a question on the baseline survey).
  Participants
    Race/Ethnicity: number analyzed (Participants) | 134 | 126 | 126 | 121 | 507
    Race/Ethnicity: Caucasian | 84 | 86 | 92 | 88 | 350
    Race/Ethnicity: Black / African | 11 | 12 | 13 | 7 | 43
    Race/Ethnicity: Hispanic / Latinx | 19 | 7 | 7 | 15 | 48
    Race/Ethnicity: All others | 20 | 21 | 14 | 11 | 66
Daily E-cigarette use, baseline [Count of Participants; unit: Participants] — Population: Missing data on one participant (due to not answering a question on the baseline survey).
  Participants
    number analyzed (Participants) | 134 | 126 | 125 | 122 | 507
    Daily E-cigarette use at baseline | 99 | 97 | 96 | 103 | 395
    Less than daily use at baseline | 35 | 29 | 29 | 19 | 112
E-cigarette use 30+ times per day [Count of Participants; unit: Participants] — Population: Missing data on 16 participants (due to not answering a question on the baseline survey).
  Participants
    number analyzed (Participants) | 132 | 121 | 120 | 119 | 492
    Use 30+ times per day | 38 | 48 | 46 | 51 | 183
    Use <30 times per day | 94 | 73 | 74 | 68 | 309

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Vaping Abstinence
Description: Self-report of no use of e-cigarettes in the past 7 days at the time of the 3-month outcome survey.
Time Frame: 3 months after the first coaching call (occurred at baseline)
Population: All participants who were fully enrolled at baseline are included. Those missing outcome data are imputed as not abstinent.
Measure: Count of Participants; unit: Participants
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Number analyzed (Participants) | 134 | 126 | 126 | 122
Participants | 55 | 54 | 61 | 59
Statistical Analysis 1: Comparison: CoachingOnlyArm vs DigitalArm vs CoachingNRTArm vs DigitalNRTArm; Comparison of NRT vs. no-NRT in model adjusted for receipt of digital component; Test type: Superiority; p = 0.14, Regression, Logistic — A priori threshold was 0.10; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.91 to 1.84] — Reported OR is NRT receipt vs. not, so values >1 indicate higher odds of abstinence among those receiving NRT
Statistical Analysis 2: Comparison: CoachingOnlyArm vs DigitalArm vs CoachingNRTArm vs DigitalNRTArm; Comparison of Digital vs. no Digital in model adjusted for receipt of NRT component; Test type: Superiority; p = 0.84, Regression, Logistic — A priori threshold was 0.10; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.73 to 1.47] — Reported OR is Digital receipt vs. not, so values >1 indicate higher odds of abstinence among those receiving the Digital component

2. Secondary Outcome: Vaping Abstinence
Description: Self-reported 30-day point prevalence vaping abstinence
Time Frame: Assessed 3 months after study enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Number analyzed (Participants) | 134 | 126 | 126 | 122
Participants | 46 | 45 | 52 | 53

3. Secondary Outcome: E-cigarette Dependence - PROMIS-E
Description: Self-reported e-cigarette dependence using the Patient Reported Outcomes Measurement Information System - E-cigarettes (PROMIS-E) questionnaire. Minimum t-score 0, maximum t-score 100. Larger scores indicate greater dependence.
Time Frame: Assessed 3 months after study enrollment
Population: Participants who were not 7 day point prevalence abstinent at the 3-month follow up survey and had complete PROMIS-E data at both baseline and the 3-month follow up survey.
Measure: Mean (Standard Deviation); unit: change in t-score
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Number analyzed (Participants) | 38 | 29 | 33 | 28
change in t-score | -5.5 (10.3) | -2.6 (7.8) | -6.5 (10.5) | -7.3 (11.0)

4. Secondary Outcome: E-cigarette Dependence - Penn State E-cigarette Dependence Index
Description: Self-reported e-cigarette dependence using the Penn State E-cigarette Dependence Index. The total score ranges from 0-20, with higher values indicating greater dependence.
Time Frame: Assessed 3 months after study enrollment
Population: Participants who were not 7-day point prevalence abstinent at the 3-month survey and completed all questions as required by the PSU dependence questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Number analyzed (Participants) | 26 | 16 | 22 | 15
Participants
  Not dependent (0-3) | 1 | 1 | 4 | 0
  Low dependence (4-8) | 10 | 1 | 5 | 3
  Medium dependence (9-12) | 8 | 3 | 9 | 3
  High dependence (13+ | 7 | 11 | 4 | 9

5. Secondary Outcome: Changes in E-cigarette Use Frequency
Description: Self-reported e-cigarette use frequency in the last 30 days. Measured at baseline and 3 months after study enrollment and calculated as the change between these two time points (3 months - baseline).
Time Frame: Assessed at baseline and 3 months after study enrollment
Population: Participants who were not 7-day point prevalence abstinent at the 3-month survey and were not missing data on number of days vaped in the past 30 on either the 3-month or baseline survey.
Measure: Mean (Standard Deviation); unit: Vaping days past month
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
Number analyzed (Participants) | 44 | 31 | 34 | 30
Vaping days past month | -7.9 (9.0) | -6.9 (9.3) | -9.3 (9.9) | -5.5 (10.0)

ADVERSE EVENTS:
Time Frame: During study participation (3 months)
Description: All-Cause Mortality and Serious Adverse Events were collected in all participants. We did not collect Other (Not Including Serious) Adverse Events on all participants, only those who completed the follow-up survey, which varied by randomized group (n=102 CoachingOnly; n=87 for DigitalArm; n=96 for CoachingNRTArm; n=94 for DigitalNRTArm)"
Arm/Group | CoachingOnlyArm | DigitalArm | CoachingNRTArm | DigitalNRTArm
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/126 | 0/126 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/126 | 0/126 | 0/122
Other Adverse Events (participants affected / at risk) | 14/102 | 10/87 | 33/96 | 33/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CoachingOnlyArm (N=102) | DigitalArm (N=87) | CoachingNRTArm (N=96) | DigitalNRTArm (N=94)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 2 | 18 | 14
Sore or dry mouth (Gastrointestinal disorders) | 2 | 2 | 10 | 9
Headache (Nervous system disorders) | 4 | 4 | 12 | 14
Dizziness (Nervous system disorders) | 3 | 2 | 6 | 8
Sleeplessness / trouble sleeping (Nervous system disorders) | 1 | 2 | 6 | 9
Bad or vivid dreams / nightmares (Psychiatric disorders) | 0 | 2 | 6 | 7
Nausea / upset stomach (Gastrointestinal disorders) | 3 | 2 | 8 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04974580/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04974580/SAP_001.pdf
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04974580/ICF_002.pdf